CLINICAL TRIAL: NCT00502424
Title: Study of the Effectiveness of a Positioning Hand Splint for Wrist, Fingers and Thumb in Patients With Arthritis Rheumatoid
Brief Title: The Effectiveness of a Nighttime Positioning Hand Splint in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2304
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2007-07-17 (Estimated); Status verified 2007-04

CONDITIONS: Rheumatoid Arthritis.
Keywords: Rheumatoid Arthritis; Hand; Splint; Occupational Therapy
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Splint

SUMMARY:
The purpose of the present study was to evaluate the effectiveness of a nighttime positioning hand splint in patients with RA in terms of pain, grip and pinch strength, upper limb function, quality of life, and patient satisfaction. The hypothesis is that the stabilization of hand during nighttime could decrease pain and consequently improve quality of life.

DETAILED DESCRIPTION:
The involvment of wrist and fingers is very common in RA and it could affect hand function and, consequently, affect activities of daily living (ADL). Some authors suggest that the rest of hand could decrease pain and inflammation. Splints are external appliances that used in a specific body part provides the best alignment and rest in correct functional position. The goal of a hand, fingers and thumb in RA is stabilize the hand while the patients are not making theirs ADL and try to decrease the pain.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis classified according to the ACR criteria.
* Use of the same remissive drugs for at least 6 months before the intervention and the same doses of the same corticosteroids and nonsteroidal anti-inflammatory drugs for at least one month before the study.
* A score ≥ 3 and ≤ 7 on a visual analog scale (VAS) for pain in the more aching hand.
* Agreement to participate in the study, and signing of a free informed consent form.

Exclusion Criteria:

* Presented deformities in the more aching hand that did not permit fabrication of the splint.
* Patients using any other type of upper limb splint.
* Patients with a surgery scheduled within 6 months after the study.
* Patients allergic to the splint material.
* Patients with mental deficiency.
* Patients who lived in inaccessible areas.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-07; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Pain using VAS at rest in cm, strength (grip and pinch), activities of daily living using HAQ questionnaire, hand function using DASH questionnaire and satisfaction with use by a likert scale of five points (much worst to much better). | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Ana Carolina R Silva, student, Principal Investigator — Federal University of São Paulo
Locations (1):
- UNIFESP - Federal University of Sao Paulo, São Paulo, São Paulo, Brazil